CLINICAL TRIAL: NCT04814485
Title: A Prospective, Single-center Clinical Study to Explore the Efficacy and Safety of SHR-1020 Combined With Albumin-bound Paclitaxel in the Second-line Treatment of Pancreatic Cancer
Brief Title: Efficacy and Safety of SHR-1020 Combined With Albumin-bound Paclitaxel in the Second-line Treatment of Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANC-2nd-IIT-FMTN-naP
Record Dates: First submitted 2021-03-17; First posted 2021-03-24 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2020-12

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1020 combined with albumin-bound paclitaxel (Experimental): SHR-1020 combined with albumin-bound paclitaxel
  Interventions: Drug: SHR-1020+albumin-bound paclitaxel

INTERVENTIONS:
Drug: SHR-1020+albumin-bound paclitaxel — SHR-1020 combined with albumin-bound paclitaxel for advanced pancreatic cancer
  Other Names: Nab-paclitaxel， Paclitaxel-albumin

SUMMARY:
This study is being conducted to explore the efficacy and safety of SHR-1020 combined with albumin-bound paclitaxel in the second-line treatment of advanced pancreatic cancer.

DETAILED DESCRIPTION:
This trial is a prospective, single-center, single-arm clinical research. Advanced pancreatic cancer is an aggressive disease with extremely low 5-year survival rate. For advanced pancreatic cancer patients who failed with first-line treatment, subsequent treatment options are limited. SHR-1020 combined with albumin-bound paclitaxel could through multiple mechanisms such as block tumor mitosis, inhibit tumor angiogenesis, inhibit interstitial fibrosis to achieve anti-tumor effect.

The safety and efficacy of this study will be assessed through ORR, DCR,PFS, OS , and adverse effects as graded by CTCAE 5.0.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed as metastatic or locally advanced unresectable pancreatic ductal adenocarcinoma by histopathology or cytology, at least one measurable lesion conforming to RECIST 1.1 criteria.
* Disease progresses or intolerance for first-line standard treatment, including patients who relapsed or metastasized within 6 months of neoadjuvant or adjuvant therapy
* ECOG score 0-2
* Adequate organ and bone marrow function
* The expected survival time is ≥ 12 weeks
* Had normal swallowing function, without dysfunction of gastrointestinal absorption
* Willing to consent and signed the informed consent, and able comply with the planned visit, research treatment, laboratory examination and other test procedures

Exclusion Criteria:

* The patient has previously received anti-angiogenic drugs or albumin-bound paclitaxel;
* The first study drug treatment was less than 2 weeks or 5 half-lives (in terms of longer) from the last chemotherapy or 5 half-lives from the last targeted therapy
* Known to be allergic to the active ingredients or excipients in this study.
* Had other active malignant tumors within 5 years before entering the study.
* Subject with cerebral metastasis
* Have a clear history of serious and uncontrolled other disease or mental disorders;
* Other chemotherapy, targeted therapy, hormonotherapy, immunotherapy, radiotherapy or traditional Chinese medicine should be used for anti-tumor therapy
* Other situations that the researcher considers inappropriate to participate in the research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
ORR (Objective Response Rate) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first,assessed up to 12 months]
  Containing the incidence of complete response (CR) and partial response (PR). Evaluated according to RECIST 1.1 criteria，subjects received their first tumor imaging evaluation at 8 weeks after the treatment start, followed by imaging evaluation every 2 cycles.

SECONDARY OUTCOMES:
DCR (Disease Control Rate) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first,assessed up to 12 months]
  Containing the incidence of complete response (CR), partial response (PR) and stable disease (SD).Evaluated according to RECIST 1.1 criteria，subjects received their first tumor imaging evaluation at 8 weeks after the treatment start, followed by imaging evaluation every 2 cycles.
PFS (Progression-Free-Survival) | From date of treatment start until the date of progression or the date of death due to any caus, assessed up to 12 months
  From date of treatment start until the date of progression or the date of death due to any cause.Evaluated according to RECIST 1.1 criteria，subjects received their first tumor imaging evaluation at 8 weeks after the treatment start, followed by imaging evaluation every 2 cycles.
6mPFS | Up to 6 months
  6-month- Progression-Free-Survival rate. Evaluated according to RECIST 1.1 criteria，subjects received their first tumor imaging evaluation at 8 weeks after the treatment start, followed by imaging evaluation every 2 cycles.
OS (overall survival) | From date of treatment start until the date of death from any cause or censored at the last day that the patient is documented to be alive, whichever came first, assessed up to 12 months
  From date of treatment start to any cause death or last follow-up.
Adverse events (per CTCAE v5.0 criteria) | Up to 12months
  To evaluate the adverse events of patients with advanced pancreatic cancer after treated with SHR-1020 plus albumin-bound paclitaxel

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No